CLINICAL TRIAL: NCT04114786
Title: MRI-based Immobilization and Planning: A Feasibility Study of a Novel Inverse Method for CNS Radiotherapy
Brief Title: 3D Printed Mask for GBM and Brain Mets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5753
Record Dates: First submitted 2019-07-25; First posted 2019-10-03 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Brain Cancer
Keywords: Radiation; Brain Cancer; Glioblastoma; 3D printed mask
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed mask (Experimental): Patients will undergo the standard CT SIM, and MR SIM necessary for radiation therapy, creating the masks from the MRIs. Prior to the start of their treatment, patients will have an additional CT scan with the 3D printed mask to confirm safety and treatment accuracy. Patients will then proceed with their standard radiation therapy, immobilized with the mask.The group will complete a mask tolerability questionnaire throughout the course of their treatment to capture the level of discomfort patients may feel with either masks.
  Interventions: Device: 3D-printed mask
- Control group (Active Comparator): Control group that will be treated with the standard thermoplastic mask, as a comparison measure. The group will complete a mask tolerability questionnaire throughout the course of their treatment to capture the level of discomfort patients may feel with either masks.
  Interventions: Device: Thermoplastic mask

INTERVENTIONS:
Device: 3D-printed mask — After patient is enrolled to the study, patients will have CT Sim. MR Sim (used to create 3D printed mask for intervention arm only) CT sim repeat (for intervention arm only) before start of radiation Patients will be asked to fill out a questionnaire after each CT Scan, and during the first and last week of radiation treatment
  Arms: 3D-printed mask
Device: Thermoplastic mask — Patients will undergo standard of care simulation, planning and treatment with conventional workflow using thermoplastic mask.They will complete the tolerability questionnaire after CT-sim, and towards the end of the first and last week of treatment.
  Arms: Control group

SUMMARY:
This is a single site, investigator initiated study that aims to explore the feasibility of using a personalized 3D printed immobilization mask for CNS patients undergoing radiation therapy.

For the purpose of this study, patients will undergo the standard CT SIM, and MR SIM necessary for radiation therapy, creating the masks from the MRIs. Prior to the start of their treatment, patients will have an additional CT scan with the 3D printed mask to confirm safety and treatment accuracy. Patients will then proceed with their standard radiation therapy, immobilized with the mask. There will be a control group that will be treated with the standard thermoplastic mask, as a comparison measure. Both groups will complete a mask tolerability questionnaire throughout the course of their treatment to capture the level of discomfort patients may feel with either masks.

DETAILED DESCRIPTION:
All patients referred for radiotherapy have had a previous diagnostic imaging study (CT-scan or more commonly MRI) showing the disease at the central nervous system (CNS). Moreover, after surgical biopsy or resection, many Centers perform repeated post-operative imaging. Despite all prior imaging, when radiotherapy treatment is decided, all patients undergo another imaging study (CT simulation [CT-sim]) in which patient's head is placed in a reproducible position, and endure a moulding procedure to create a personalized plastic mask for securing the patient's head in a fixed position during the CT acquisition, and reproduced at the subsequent radiation treatment sessions. Typical wait times between moulding, CT-sim and the first radiation treatment is 3-7 days. If a method would be available to accurately recreate the patient's position during diagnostic imaging and reproduce it during radiation treatments without the need for a moulding session or CT-sim, the treatment process can be streamlined and wait times shortened for patients.

Previous studies using 3D printing technology in radiotherapy (such as brachytherapy applicators) have shown that these employed materials are safe for use in clinical settings, and 3D printers can accurately produce devices of various shapes and sizes for clinical use.

In this study, we propose a novel workflow in which patient's position at diagnostic imaging is reproduced with a 3D-printed patient-specific immobilization device, enabling the use of the same diagnostic imaging for planning purposes in lieu of dedicated simulation and moulding sessions, to decrease wait times for patients between diagnostic imaging and start of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patient with high-grade glioma considered for external beam radiotherapy (15 fractions or more) with or without Temozolamide, or patients with brain metastases considered for fractionated LINAC-based external beam radiotherapy (5 fractions or more) as primary or adjuvant treatment.
* No contraindications to MRI
* No other medical conditions deemed by the PI to make patient ineligible for the study (i.e. claustrophobia, confusion, delirium).

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Treatment planning time | Baseline to week 1
  Overall treatment planning time: from planning MRI acquisition to first treatment session delivery.
3D-mask confection time | Baseline to week 1
  3D-mask confection time during radiation therapy
Inter- and intra-fraction motion | Baseline to week one
  Inter- and intra-fraction motion during radiation therapy
Patient reported adverse events and tolerability of mask | First scan through to end of radiation treatment, an average 8 weeks
  CT-simulation, first and last week of radiation treatment

SECONDARY OUTCOMES:
Gamma values and histograms for MRI-based plans | First scan through to end of radiation treatment, an average 8 weeks
  Gamma values and histograms for MRI-based plans of Planning MRI and Radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Berlin, <D, Principal Investigator — Princess Margaret
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No